CLINICAL TRIAL: NCT04300270
Title: Validation of a Novel Smartphone-based Photoplethysmographic Method for Ambulatory Heart Rhythm Monitoring in Connection to Treatment of Atrial Fibrillation With Direct Current Cardioversion
Brief Title: Validation of a Novel Smartphone-based Method for Heart Rhythm Monitoring in the Home Environment
Status: Active, not recruiting | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: Danderyd Hospital (Other)
Responsible Party: Principal Investigator, Johan Engdahl, Associate Professor, Karolinska Institutet
Other Study IDs: SmartBeats
Record Dates: First submitted 2020-03-04; First posted 2020-03-09 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Atrial Fibrillation; Atrial Flutter; Arrhythmia
Keywords: Smartphone; Photoplethysmography; Cardioversion; Telemonitoring; Validation; Mobile ECG
MeSH Terms: conditions — Atrial Fibrillation; Atrial Flutter; Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Validation cohort: Participants in validation of the novel smartphone-based photoplethysmographic method for ambulatory heart rhythm diagnostics.
  Interventions: Device: Smartphone PPG recordings; Device: Smartphone ECG
- Clinical implementation cohort: Participants in a clinical implementation of the novel smartphone-based photoplethysmographic method for ambulatory heart rhythm diagnostics.
  Interventions: Device: Smartphone PPG recordings; Device: Smartphone ECG

INTERVENTIONS:
Device: Smartphone PPG recordings — Smartphone camera PPG recordings using a novel software application.
Device: Smartphone ECG — Smartphone connected one-lead ECG recordings.
  Other Names: Alivecor Kardia Mobile ECG

SUMMARY:
Atrial fibrillation is a heart rhythm disorder with increased risk of stroke, heart failure, dementia and death. The severity of symptoms in atrial fibrillation varies markedly, ranging from no symptoms to those with disabling symptoms. An ECG recording is currently mandatory for diagnosing atrial fibrillation. A portable method for heart rhythm diagnostics that is readily available is currently missing in clinical practice. If a standard smartphone could be used for heart rhythm diagnostics, the availability could improve greatly.

Treatment with direct current cardioversion is a procedure in which the heart rhythm is normalized by an electrical shock through the chest. Patients with atrial fibrillation are in some cases recommended treatment with direct current cardioversion but the procedure is costly, has a high recurrence rate and includes an increased risk for stroke. In this study we will validate the use of a novel smartphone-based method for heart rhythm diagnostics when used by patients in their home environment. The novel method is using the smartphone camera as a sensor. Patients will be doing heart rhythm measurements with the novel smartphone-based method in their home environment for 30 days after successfully receiving treatment of atrial fibrillation with direct current cardioversion. The novel smartphone-based method will be validated against simultaneous recordings with mobile ECG.

We will also study the feasibility in using smartphone recordings and mobile ECG in the home environment the weeks before receiving treatment with direct current cardioversion, to study the possible benefit of detecting spontaneous conversions to normal heart rhythm and missed doses of treatment with blood thinning medication, both of which will lead to cancellation or detention of the cardioversion procedure.

DETAILED DESCRIPTION:
Atrial fibrillation is a heart rhythm disorder with increased risk of stroke, heart failure, dementia and death. The severity of symptoms in atrial fibrillation varies markedly, ranging from no symptoms to those with disabling symptoms. An ECG recording is currently mandatory for diagnosing atrial fibrillation.

The availability of long-term ECG and portable ECG registration for heart rhythm diagnostics within the healthcare sector is severely limited by waiting time both for ECG recording and for analysis and reporting. A method for heart rhythm diagnostics that is readily available is currently lacking in clinical practice, except for hospitalization, which is very costly and has low availability.

The lack of a method for diagnosis of heart rhythm disorders and atrial fibrillation that is readily available, cost-effective and simple to use is a problem for both the patients and for the healthcare system as a whole. The limited availability of patient-related diagnostics thus means that many patients, even those with symptoms, remain undiagnosed and thus untreated, which in turn means that the missing diagnosis gives an increased risk of stroke. If a standard smartphone could be used for reliable heart rhythm diagnostics, the availability could improve greatly.

Treatment with direct current cardioversion is a procedure in which the heart rhythm is normalized by an electrical shock through the chest. Patients with atrial fibrillation could in some cases be treated with cardioversion but the procedure is costly, has a high recurrence rate and includes an increased risk for thromboembolism and stroke. The benefit of the treatment is mainly symptomatic, with no proven long-term effects of mortality or morbidity.

In this study we will validate the use of a novel smartphone-based method for heart rhythm diagnostics when used by patients in their home environment after receiving treatment with direct current cardioversion. The novel method is using the smartphone camera as a sensor and records photoplethysmographic (PPG) measurements. We will also study the feasibility in using smartphone and mobile ECG recordings peri-cardioversion, to study the possible benefit of detecting pre-cardioversion spontaneous conversions to sinus rhythm and non-adherence to treatment with oral anticoagulants, both of which will lead to cancellation or detention of the cardioversion procedure. We will also detect the timing of post-cardioversion early recurrences into atrial fibrillation, as well as the heart rate and symptoms associated to recurrence, if any.

The objective of this study is to:

1. Validate heart rhythm measurements registered with a novel smartphone-based method using PPG-measurement technology compared to mobile ECG technology in patients with atrial fibrillation. The validation involves evaluating whether PPG-measurement technology using a novel smartphone-based method provides sufficient diagnostic performance in the home environment / outpatient environment compared to outpatient mobile ECG measurements.
2. Study if pre-cardioversion heart rhythm recordings will reduce the number of same day cancellations of treatment of atrial fibrillation with planned direct current cardioversion.

For the validation part, patients who visit the cardiac day care department at the department of Cardiology, Danderyd University Hospital, for treatment with outpatient direct current cardioversion of atrial fibrillation or atrial flutter are asked about participating by physicians or research nurses. Each patient will prior to inclusion in the study be given full and adequate verbal and written information regarding the objective and procedures of the study and possible risks involved. Written consent is obtained from the physician or research nurse.

A 60-second heart rhythm measurement using a smartphone is recorded before the patient receives treatment with direct current cardioversion. The smartphone used is the same device that the patient will be using in their home for 30 days after the treatment. The measurement includes PPG-measurement from the camera of the smartphone as well as a simultaneous one lead ECG-registration done with a small ECG-device attached to the back of the smartphone.

The patient is interviewed about their medical history and their current symptoms. If the treatment is successful and the patient's heart rhythm is converted back to normal sinus rhythm, the patient is included in the study. The patient's heart rhythm is verified with an ECG measurement recorded approximately one hour after the cardioversion treatment.

When the patients are discharged from the hospital they are given a smartphone that they will be recording simultaneous PPG- and ECG-recordings with, at least twice daily for a period of 30 days post-cardioversion in their home.

For the clinical implementation part, patients scheduled for direct current cardioversion at Danderyd University Hospital will be included at least 2 weeks prior to the scheduled treatment. Information regarding co-morbidities, echocardiographic parameters and current medication will be collected from interviews and medical records.

All individuals scheduled for direct current cardioversion will be invited to a screening visit and asked to sign a written consent form. After consent, their heart rhythm will be recorded and those with sinus rhythm will be excluded. Participants with atrial fibrillation or atrial flutter will be randomized 1:1 to pre-cardioversion heart rhythm monitoring, or no monitoring pre-cardioversion.

Participants randomized to active pre-cardioversion rhythm monitoring (intervention group) will be instructed in the use of smartphone rhythm recordings (using simultaneous PPG and mobile ECG). They will be recording both their heart rhythm and oral anticoagulant treatment adherence with the same smartphone application. This information will give the investigators the possibility to cancel or postpone the scheduled cardioversion visit in advance for those with spontaneous rhythm conversion to sinus rhythm and for those with non-adherence to oral anticoagulant treatment.

Participants randomized to passive pre-cardioversion rhythm monitoring (control group) will be instructed in the use of smartphone rhythm recordings (using simultaneous PPG and mobile ECG). The control group will be recording only heart rhythm and not treatment adherence. The heart rhythm recordings made in the control group will be reviewed after the participants treatment with direct current cardioversion.

After the treatment with direct current cardioversion, all participants are followed up in one common cohort.

ELIGIBILITY:
Validation cohort:

Inclusion Criteria:

* Patients undergoing direct current cardioversion successfully for treatment of atrial fibrillation or atrial flutter and have a normal heart rhythm after the treatment.

Exclusion Criteria:

* Patients with implantable cardiac devices.

Clinical implementation cohort:

Inclusion Criteria:

* Patients planned for direct current cardioversion for treatment of atrial fibrillation or atrial flutter.

Exclusion Criteria:

* Patients with implantable cardiac devices.
* Patients with a spontaneous return to sinus rhythm diagnosed at a screening visit 2 to 4 weeks prior to the scheduled treatment with direct current cardioversion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing direct current cardioversion for treatment of atrial fibrillation or atrial flutter at Danderyd University Hospital.
Sampling Method: Probability Sample
Enrollment: 480 (Estimated)
Dates: Start 2018-11-27 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Performance of the novel smartphone-based photoplethysmographic method for heart rhythm diagnostics and discrimination of atrial fibrillation from normal heart rhythm. | Daily measurements during 30 days
  Sensitivity, specificity, positive predictive value, negative predictive value, receiver operating characteristic (ROC) curve analysis.

SECONDARY OUTCOMES:
Independent predictors for recurrence of atrial fibrillation within 30 days of treatment with direct current cardioversion. | 30 days
  Odds ratio
Predictors for recurrence of atrial fibrillation within 30 days of treatment with direct current cardioversion using deep learning and machine learning techniques. | 30 days
Participant compliance for recording heart rhythm with the novel smartphone-based method twice daily for 30 days. | 30 days
  Actual compared to expected number of recordings. Proportion of recordings with interpretable signal quality.
Correlation between patient self-reported symptoms and recorded heart rhythm. | 30 days
  Correlation between heart rhythm perceived by the participant (dichotomized into sinus rhythm or atrial fibrillation) and actual rhythm recorded on handheld ECG (dichotomized in the same way), expressed as correlation coefficient R and cohen´s kappa.
Proportion of same day cancellations for planned treatment of atrial fibrillation with cardioversion for patients using the novel smartphone-based photoplethysmographic method for heart rhythm monitoring prior to the treatment compared to no monitoring. | 2 to 4 weeks
  Comparison of proportions

CONTACTS AND LOCATIONS:
Overall Officials: Johan Engdahl, Principal Investigator — Karolinska Institutet
Locations (1):
- Danderyd University Hospital, Stockholm, Sweden

REFERENCES:
- [Derived] Fernstad J, Svennberg E, Aberg P, Kemp Gudmundsdottir K, Jansson A, Engdahl J. External validation of a machine learning-based classification algorithm for ambulatory heart rhythm diagnostics in pericardioversion atrial fibrillation patients using smartphone photoplethysmography: the SMARTBEATS-ALGO study. Europace. 2025 Mar 28;27(4):euaf031. doi: 10.1093/europace/euaf031. PMID 39960451